CLINICAL TRIAL: NCT00545701
Title: Immunogenicity and Safety of an Intramuscular A/H5N1 Inactivated, Split Virion Pandemic Influenza Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GPA11
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; A/H5N1 strain; Orthomyxoviridae Infections; Influenza Pandemics
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: A/H5N1 inactivated, split-virion influenza virus

INTERVENTIONS:
Biological: A/H5N1 inactivated, split-virion influenza virus — 0.5 mL, Intramuscular

SUMMARY:
The trial is a Phase II, open-label trial in healthy subjects aged 18 to 60 years to support the immunogenicity data from previous clinical studies.

Objectives:

* To describe the immune response 21 days after each vaccination.
* To describe the safety profiles following each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 60 years on day of inclusion.
* Informed Consent Form signed.
* Able to attend all scheduled visits and to comply with all trial procedures.
* For a woman, inability to bear a child or negative urine pregnancy test.
* For a woman of child-bearing potential, use of an effective method of contraception or abstinence for at least 4 weeks prior to and at least 4 weeks after each vaccination.

Exclusion Criteria:

* Systemic hypersensitivity to any component of the vaccine or a life-threatening reaction after previous administration of a vaccine containing the same substances (egg proteins, chick proteins, thimerosal, aluminum, neomycin, formaldehyde, and octoxinol 9).
* Febrile illness (oral temperature >= 37.5°C) on the day of inclusion.
* Breast-feeding.
* Previous vaccination with an avian flu vaccine.
* Participation in a clinical trial (drug, device, or medical procedure) within 4 weeks prior to the first vaccination.
* Planned participation in another clinical trial during the present trial period.
* Congenital or acquired immunodeficiency, or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy.
* Chronic illness that could interfere with trial conduct or completion (e.g. cardiac, renal, diabetes, or auto-immune disorders).
* Current alcohol or drug abuse that may interfere with the subject's ability to comply with trial procedures.
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with the assessment of immune response.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of A/H5N1 inactivated, split-virion influenza virus vaccine | Day 42 post-vaccination 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (2):
- Australia (2):
  - Adelaide
  - Queensland

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com